CLINICAL TRIAL: NCT06598462
Title: A Phase 2, Randomized, Double-Blind, Multicenter, Placebo Controlled Study With an Extension to Investigate the Efficacy and Safety of NSI-8226 in Adults With Eosinophilic Esophagitis (ALAMERE)
Brief Title: A Study to Investigate the Efficacy and Safety of NSI-8226 in Adults With Eosinophilic Esophagitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uniquity One (UNI) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSI-8226-201
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Solrikitug low dose (Experimental): Solrikitug
  Interventions: Biological: Solrikitug Low Dose
- Solrikitug mid dose (Experimental): Solrikitug
  Interventions: Biological: Solrikitug Mid Dose
- Solrikitug high dose (Experimental): Solrikitug
  Interventions: Biological: Solrikitug High Dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Solrikitug Low Dose — Solrikitug low dose subcutaneous injection
  Arms: Solrikitug low dose
Biological: Solrikitug Mid Dose — Solrikitug mid dose subcutaneous injection
  Arms: Solrikitug mid dose
Biological: Solrikitug High Dose — Solrikitug high dose subcutaneous injection
  Arms: Solrikitug high dose
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
Phase 2 study to evaluate the safety, tolerability, PK, immunogenicity, and pharmacodynamics of solrikitug in adult participants with eosinophilic esophagitis.

DETAILED DESCRIPTION:
This is a 24-week randomized, double-blind, placebo-controlled Phase 2 clinical study with a 28-week extension to evaluate the safety, tolerability, PK, immunogenicity, and pharmacodynamics of 3 dose levels of solrikitug versus placebo on top of standard of care in adult participants with EoE.

Approximately 180 adult participants with EoE will be randomized at approximately 80 sites. Participants will receive solrikitug, or placebo, administered via subcutaneous injection at the study site, over a 24-week treatment period followed by a 28-week extension period. The study also includes a post-treatment follow-up period of 16 weeks.

ELIGIBILITY:
Key inclusion criteria

Part A

* Participant must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
* Established diagnosis of EoE with a previous EGD and esophageal biopsy confirming diagnosis of EoE.
* Participants who have symptomatic EoE as defined by a history of on average at least 2 episodes of dysphagia per week in the 4 weeks prior to Screening.
* Must remain on a stabilized diet for at least 8 weeks prior to Visit 1 and during the course of the study.
* May be on any background PPI and/or STC, during the course of the study, as long as background medications have been stable for at least 8 weeks prior to the Screening and must agree to no changes to background medication or dosage unless medically indicated.
* Discontinuation of any marketed investigational drug or biologic (monoclonal or polyclonal antibody) within 30 days or 5 half-lives prior to screening, whichever is longer.
* Participants should have previously documented standard of care treatment, which could include PPI and/or STC and/or diet.

Key exclusion criteria

Part A

* Female participant who is pregnant or breastfeeding.
* Have a history or presence of any other gastrointestinal disorders such as active Helicobacter pylori infection, history of achalasia, hyper eosinophilic syndrome and eosinophilic granulomatosis with polyangiitis, esophageal varices, Crohn's disease, ulcerative colitis, inflammatory bowel disease, celiac disease, eosinophilic enteritis, gastritis, colitis, diverticulitis, irritable bowel syndrome, or other clinically significant gastrointestinal conditions as per Investigator discretion.
* Esophageal stricture that prevents the easy passage of a standard endoscope or any critical esophageal stricture that requires dilation at screening.
* Esophageal dilation performed within 8 weeks prior to screening.
* Participant has a known hypersensitivity to any component of the formulation of solrikitug, including any of the excipients, or a history of anaphylactic reaction to any therapeutic monoclonal antibody.

Part B

* Participants who, during Part A, developed a serious adverse event (SAE) and/or adverse event (AE) deemed related to study drug, which in the opinion of the investigator could indicate that continued treatment with study drug may present and unreasonable risk to the participant.
* Participants who became pregnant during Part A.
* Participants who are prematurely discontinued from study drug due to AE (patients who are prematurely discontinued from study drug due to lack of efficacy are eligible to enter Part B).
* Patients who did not undergo endoscopy with biopsies prior to receiving rescue treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Histological response of peak esophageal eosinophil per HPF count of ≤6 | Week 24
Change from baseline in DSQ (Dysphagia Symptom Questionnaire) score | Week 24
  The DSQ score is calculated over 14-day period and ranges from 0 to 84, with a lower score indicating less severe dysphagia.

SECONDARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) | To Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Lee, MD, Study Chair — Vice President, Clinical Research
Locations (55):
- United States (32):
  - Research Site 1039, Dothan, Alabama
  - Research Site 1037, Paradise Valley, Arizona
  - Research Site 1018, Peoria, Arizona
  - Research Site 1037, Scottsdale, Arizona
  - Research Site 1003, Tucson, Arizona
  - Research Site 1023, Englewood, California
  - Research Site 1015, San Diego, California
  - Research Site 1027, Bristol, Connecticut
  - Research Site 1027, Cromwell, Connecticut
  - Research Site 1040, Inverness, Florida
  - Research Site 1001, Jacksonville, Florida
  - Research Site 1007, Boise, Idaho
  - Research Site 1048, Glenview, Illinois
  - Research Site 1048, Gurnee, Illinois
  - Research Site 1022, Iowa City, Iowa
  - Research Site 1033, Topeka, Kansas
  - Research Site 1032, Chevy Chase, Maryland
  - Research Site 1004, Boston, Massachusetts
  - Research Site 1013, Wyoming, Michigan
  - Research Site 1006, Plymouth, Minnesota
  - Research Site 1016, Reno, Nevada
  - Research Site 1045, Freehold, New Jersey
  - Research Site 1043, Jackson, New Jersey
  - Research Site 1026, Chapel Hill, North Carolina
  - Research Site 1021, High Point, North Carolina
  - Research Site 1012, Columbus, Ohio
  - Research Site 1020, Harrisburg, Pennsylvania
  - Research Site 1014, Dallas, Texas
  - Research Site 1008, Houston, Texas
  - Research Site 1036, Pearland, Texas
  - Research Site 1002, Ogden, Utah
  - Research Site 1017, Sandy City, Utah
- Australia (9):
  - Research Site 1108, Newcastle, New South Wales
  - Research Site 1110, Maroochydore, Queensland
  - Research Site 1103, South Brisbane, Queensland
  - Research Site 1107, Woolloongabba, Queensland
  - Research Site 1106, Box Hill, Victoria
  - Research Site 1102, Fitzroy, Victoria
  - Research Site 1109, Murdoch, Western AUS
  - Research Site 1111, Maroochydore
  - Research Site 1107, Woolloongabba
- Belgium (2):
  - Research Site 1152, Bruges
  - Research Site 1153, Tournai
- Research Site 1258, Verona, Italy
- Poland (7):
  - Research Site 1207, Lodz
  - Research Site 1202, Szczecin
  - Research Site 1205, Tychy
  - Research Site 1203, Warsaw
  - Research Site 1206, Warsaw
  - Research Site 1204, Warsaw
  - Research Site 1201, Warsaw
- Spain (3):
  - Research Site 1354, Barcelona
  - Research Site 1353, Madrid
  - Research Site 1351, Tomelloso
- Research Site 1551, Whitechapel, London, United Kingdom